CLINICAL TRIAL: NCT01181440
Title: A Prospective, Multicenter, Randomized, Single-Blind Clinical Investigation of Dermagraft(R) in Patients With Plantar Diabetic Foot Ulcers
Brief Title: Dermagraft(R) for the Treatment of Patients With Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABH-DG-04-04-0694
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer; Randomized trial; Clinical trial; Dermagraft; Conventional care
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

ARMS (2):
- Dermagraft(R) and conventional care (Experimental)
  Interventions: Device: Dermagraft(R)
- Conventional care only (Other)
  Interventions: Other: Conventional care

INTERVENTIONS:
Device: Dermagraft(R) — Weekly application of Dermagraft(R) with conventional care
  Other Names: human fibroblast derived dermal substitute
  Arms: Dermagraft(R) and conventional care
Other: Conventional care — Weekly application of conventional care
  Other Names: standard of care, off-loading, surgical debridement, wet-to-moist dressing
  Arms: Conventional care only

SUMMARY:
This study randomly assigns patients with plantar diabetic foot ulcers to receive conventional therapy (debridement, infection control, saline-moistened gauze dressings, and standardized off-weighting) alone or conventional therapy plus Dermagraft(R). Dermagraft is a device containing live human fibroblasts grown on an absorbable polyglactin (Vicryl) mesh. Patients are evaluated weekly until Week 12, then every four weeks until Week 32.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years old or older.
* Patient has a current diagnosis of NIDDM or IDDM.
* Patient's ulcer is present for a minimum of two weeks under the current Investigator's care
* The study ulcer has healed <50% in size during the two weeks leading up to randomization
* The study ulcer is on the plantar surface of the forefoot
* The ulcer is >/= 1.0 cm2 at Day 0 (the day of randomization).
* The ulcer extends through the dermis and into subcutaneous tissue but without exposure of muscle, tendon, bone, or joint capsule.
* The ulcer is free of necrotic debris and clinical infection and is comprised of healthy, vascular tissue and is suitable for skin grafting.
* The patient's Ankle-Arn Index by Doppler is >0.1
* There is adequate circulation to the foot to allow for healing.
* The patient's diabetes is under control as determined by the Investigator.
* Female patients capable of bearing children must test negative for pregnancy and must use an acceptable means of birth control.
* Patient and caregiver are willing to participate in the clinical study and can comply with the follow-up regimen.
* Patient or his/her legal representative has read and signed the Institutional Review Board (IRB) approved Informed Consent form.

Exclusion Criteria:

* Patient has clinical evidence of gangrene on any part of the affected foot.
* The ulcer is over a Charcot deformity.
* The ulcer has a nondiabetic etiology.
* The ulcer has tunnels or sinus tracts that cannot be completely debrided.
* The patient's diabetes is uncontrolled and could interfere with the completion of the study.
* There is a medical condition(s) that in the Investigator's opinion make the patient an inappropriate candidate for this study.
* Patient has/had a malignant disease not in remission for 5 years or more.
* Patient has acute or chronic hepatitis, cirrhosis, has a serum albumin of <2.0 gms/dL, or has alkaline phosphatase or LDH at twice the upper limit of the normal range.
* Patient is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents, or is anticipated to require such agents during the course of the study.
* Patient has Acquired Immunodeficiency Syndrome (AIDS) or is infected with Human Immunodeficiency Virus (HIV).
* Patient has participated in another study utilizing an investigational drug or device within the previous 30 days.
* The ulcer has cellulitis, osteomyelitis, or other clinical evidence of infection.
* Patient has any condition(s) which seriously compromises their ability to complete this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 1994-09; Primary Completion 1997-01 (Actual); Study Completion 1997-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete wound closure | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients with complete wound closure | 32 weeks
Time to reach 25%,50%,75%, and 100% of wound closure | 32 weeks
Percent of wound healed | 12 and 32 weeks
Wound characterization | 32 weeks
Recurrence of the ulcer | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Pollak, DPM, Principal Investigator — San Antonio Podiatry Associates, San Antonio, TX
Locations (1):
- Richard Pollak, DPM, San Antonio, Texas, United States

REFERENCES:
- [Background] Naughton G, Mansbridge J, Gentzkow G. A metabolically active human dermal replacement for the treatment of diabetic foot ulcers. Artif Organs. 1997 Nov;21(11):1203-10. doi: 10.1111/j.1525-1594.1997.tb00476.x. PMID 9384327
- [Result] Gentzkow GD, Jensen JL, Pollak RA, Kroeker RO, Lerner JM, Lerner M, Iwasaki SD, the Dermagraft Diabetic Ulcer Study Group. Improved healing of diabetic foot ulcers after grafting with a living human dermal replacement. Wounds. 1999;11:77-84